CLINICAL TRIAL: NCT01709344
Title: A Phase I Randomized Controlled Trial of a Problem-solving Occupational Therapy Intervention for Older Adult Cancer Survivors
Brief Title: Reducing Disability in Older Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Kathleen Lyons, Research Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: D12110
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PS-OT (Experimental): Problem-solving Occupational Therapy
  Interventions: Behavioral: PS-OT
- Usual care (Other): Access to all supportive and rehabilitative services available at DHMC
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: PS-OT
  Other Names: Problem-solving Occupational Therapy
  Arms: PS-OT
Other: Usual care — Supportive and rehabilitation services available at DHMC
  Arms: Usual care

SUMMARY:
Older adults who are treated for cancer are at risk of developing disabilities due to the symptoms of cancer and the side effects of treatment. Disability occurs when a person has trouble performing the activities he or she needs to do in everyday life. For example, fatigue and pain can make it difficult for an older adult to do housework, leisure, or volunteer activities. Disability makes it harder for older adults to stay active and be productive members of the community, and it can increase the costs of healthcare.

Current approaches to cancer rehabilitation focus on using exercise, education, and social support to reduce cancer treatment side effects. These are important strategies to reduce disability, yet some side effects persist despite best efforts to resolve them. To fully reduce disability, people often need to adapt their activities or the environments in which they are performed.

The goal of this study is to test an occupational therapy (OT) intervention that teaches activity planning skills to foster survivors' ability to adapt activities, routines, and environments in order to minimize disability. The project targets adults over the age of 65 who are experiencing disability during or after cancer treatment. The project has two stages. First, twelve older adult cancer survivors will individually participate in the community-based intervention. After they have completed the program the investigators will revise the intervention to emphasize what they found most effective and helpful, and to eliminate aspects of the intervention that are perceived as unhelpful or redundant. The research question for this first stage of the project is, "To what degree is it feasible for survivors to enroll in the study, complete the six-week intervention, and complete the three outcome assessments?" In the second stage of the project, the investigators will test the revised intervention, comparing it to conventional care. The research question for the second stage of the project is, "Do the people receiving the intervention have higher activity levels, greater behavioral activation, lower levels of disability, and better quality of life compared to those people who receive traditional cancer care?" The intervention is appropriate for people who have been diagnosed with any type of cancer. It is designed to focus on whatever activities are most important to each participant. The novelty of the proposed intervention lies in the combination of the OT strategies of activity and environmental adaptation with explicit training in activity planning to teach survivors to find creative ways to engage in valued activities (e.g., taking care of one's home and family members, and participating in leisure, community, social and work activities). If the intervention is effective in reducing disability, it will give us another tool to reduce the impact of cancer on the daily lives of cancer survivors.

ELIGIBILITY:
Inclusion Criteria

1. Age 65 years or older.
2. Experiencing disability as indicated by a score of > 3 on the Vulnerable Elders Survey or an answer of "yes" to the question "Do health problems interfere with your ability to carry out your social or day to day activities?"
3. Either: a. Diagnosed with any solid or hematological cancer, undergoing treatment for curative intent or within six months of completion of therapy with absence of disease recurrence; or b.Diagnosed with metastatic breast cancer or chronic hematologic malignancies with a life expectancy of > 2 years

Exclusion Criteria

1. Moderate or worse cognitive impairment as indicated by a score of 3 or less on the Callahan six-item cognitive screening tool.
2. Medical record documentation of severe mental illness (i.e., schizophrenia or bipolar disorder), active suicidal ideation, or active substance use disorder.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Disability | Eight weeks
  Late-Life Function and Disability Instrument

SECONDARY OUTCOMES:
Quality of Life | Eight weeks
  Functional Assessment of Cancer Therapy
Activity level | Eight weeks
  Activity Card Sort
Behavioral activation | Eight weeks
  Behavioral activation scale

OTHER OUTCOMES:
Depression | Eight weeks
  Patient Health Questionnaire-9 (PHQ-9)

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Lyons KD, Newman R, Adachi-Mejia AM, Whipple J, Hegel MT. Content Analysis of a Participant-Directed Intervention to Optimize Activity Engagement of Older Adult Cancer Survivors. OTJR (Thorofare N J). 2018 Jan;38(1):38-45. doi: 10.1177/1539449217730356. Epub 2017 Sep 20. PMID 28929925